CLINICAL TRIAL: NCT04262388
Title: A Multi-Cancer, Multi-State, Platform Study of Durvalumab (MEDI4736) and Oleclumab (MEDI9447) in Pancreatic Adenocarcinoma, Non-Small Cell Lung Cancer and Squamous Cell Carcinoma of the Head and Neck to Correlate Clinical, Molecular and Immunologic Parameters With DNA Methylation (DOME)
Brief Title: A Multi-Cancer, Multi-State, Platform Study of Durvalumab (MEDI4736) and Oleclumab (MEDI9447) in Pancreatic Adenocarcinoma, Non-Small Cell Lung Cancer and Squamous Cell Carcinoma of the Head and Neck to Correlate Clinical, Molecular and Immunologic Parameters With DNA Methylation
Acronym: DOME
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Overall clinical activity (ORR) for oleclumab + durvalumab is minimal across tumor types and does not support further evaluation of this doublet.
Sponsor: University Health Network, Toronto (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DOME; 19-6280 (Other: University Health Network)
Record Dates: First submitted 2020-02-05; First posted 2020-02-10 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Pancreatic Ductal Adenocarcinoma; Non-small Cell Lung Cancer; Squamous Cell Carcinoma of Head and Neck
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Squamous Cell Carcinoma of Head and Neck | interventions — durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Window (Experimental): Within each cancer type, 40 patients will be enrolled (for a total of 120 patients on study): 20 patients will be enrolled with locally advanced disease ("window") and treated with durvalumab 1500 mg given by IV x 1 dose and oleclumab 3000 mg x 2 doses every 2 weeks prior to definitive therapy (e.g. surgery).
  Interventions: Biological: Durvalumab; Biological: Oleclumab
- Metastatic (Experimental): Within each cancer type, 40 patients will be enrolled (for a total of 120 patients on study): 20 patients will be enrolled with recurrent/metastatic ("metastatic") disease and treated with durvalumab 1500 mg given by IV every 4 weeks and oleclumab 3000 mg given by IV every 2 weeks x 4 doses then IV every 4 weeks till disease progression, toxicity, withdrawal of subject consent, or another discontinuation reason.
  Interventions: Biological: Durvalumab; Biological: Oleclumab

INTERVENTIONS:
Biological: Durvalumab — Durvalumab is a human immunoglobulin G (IgG)1 kappa monoclonal antibody directed against human PD-L1. Durvalumab selectively binds human PD-L1 with high affinity and blocks its ability to bind to PD-1 and cluster of differentiation (CD)80. The fragment crystallizable (Fc) domain of durvalumab contains a triple mutation in the constant domain of the IgG1 heavy chain that reduces binding to the complement component C1q and the Fc gamma receptors responsible for mediating antibody dependent cell mediated cytotoxicity.
  Other Names: IMFINZI
Biological: Oleclumab — Oleclumab is a human immunoglobulin G1 lambda monoclonal antibody (mAb) with a triple mutation in the heavy chain constant region for reduced effector function. Oleclumab selectively binds to cluster of differentiation 73 (ecto-5'-nucleotidase) (CD73) and inhibits CD73-associated ectonucleotidase activity, thereby inhibiting the CD73-mediated production of immunosuppressive adenosine. Extracellular adenosine contributes to the immunosuppressive effects of both regulatory T cells and myeloid derived suppressor cells, among others. This, in turn, leads to increased antitumor immunity.

SUMMARY:
This is a phase II, single center, open label, multi-cohort platform study to identify a signature in tumor tissues, blood or stool that might help identify participants who are more likely to experience tumor shrinkage or side effects from the combination of the study drugs durvalumab and oleclumab. In addition, this study will see if participants with certain types of advanced cancer benefit from the experimental drug combination of durvalumab and oleclumab, will evaluate the safety and tolerability of durvalumab and oleclumab, and to understand the effects that durvalumab and oleclumab have at a molecular level in tumor cells and their effects on the immune system. This study will look at subjects with locally advanced or recurrent/metastatic pancreatic ductal adenocarcinoma (PDAC), non-small-cell carcinoma (NSCLC) and squamous cell carcinoma of head and neck (SCCHN).

Within each cancer type, 40 patients will be enrolled (for a total of 120 patients on study): 20 patients will be enrolled with locally advanced disease ("window") and treated with durvalumab 1500 mg given by IV x 1 dose and oleclumab 3000 mg x 2 doses every 2 weeks prior to definitive therapy (e.g. surgery), and 20 patients will be enrolled with recurrent/metastatic ("metastatic") disease and treated with durvalumab 1500 mg given by IV every 4 weeks and oleclumab 3000 mg given by IV every 2 weeks x 4 doses then IV every 4 weeks till disease progression, toxicity, withdrawal of subject consent, or another discontinuation reason. For locally advanced PDAC patients, approximately 10 of the 20 subjects may receive 6-8 cycles of modified FOLFIRINOX (mFFX) prior to the administration of durvalumab and oleclumab.

DETAILED DESCRIPTION:
The study hypothesis is that the combination of oleclumab (anti-cluster of differentiation [CD]73) with durvalumab (anti programmed cell death ligand 1 [PD-L1]) will demonstrate adequate safety, tolerability, and antitumor activity in subjects with locally advanced or recurrent/metastatic: pancreatic ductal adenocarcinoma (PDAC), non-small-cell lung cancer (NSCLC) and squamous cell carcinoma of head and neck (SCCHN), and that circulating free methylated DNA immunoprecipitation and high-throughput sequencing (cfMeDIP-seq) can yield cancer type-agnostic predictive biomarker(s) of response and/or toxicity in subjects receiving this combination.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years at the time of screening or age of consent
2. Written informed consent and any locally required authorization (eg, data privacy) obtained from the subject prior to performing any protocol-related procedures, including screening evaluations
3. ECOG of 0 or 1
4. Weight ≥ 35 kg
5. Must have a life expectancy of at least 12 weeeks
6. Histological or cytological confirmation
7. At least 1 measurable lesion according to RECIST version 1.1
8. Archival tumor formalin-fixed, paraffin-embedded (FFPE) specimens for correlative biomarker studies are required (1 H&E and 15 unstained slides) unless no such sample is available or insufficient sample exists. Subjects with insufficient archived tumor samples are still eligible
9. Adequate organ and marrow function
10. Females of childbearing potential who are sexually active with a nonsterilized male partner must use at least one highly effective method of contraception from screening to 180 days after the final dose of study treatment
11. Nonsterilized male subjects who are sexually active with a female partner of childbearing potential must use a male condom with spermicide from screening to 180 days after receipt of the final dose of study treatment

Exclusion Criteria:

1. Receipt of any conventional or investigational anticancer therapy within 21 days or palliative radiotherapy within 14 days prior to the scheduled first dose of study treatment.
2. Prior receipt of any immune-mediated therapy
3. Concurrent enrollment in another therapeutic clinical study. Enrollment in observational studies will be allowed
4. Any toxicity (excluding alopecia) from prior standard therapy that has not been completely resolved to baseline at the time of consent
5. Subjects with a history of Grade 3 or greater thromboembolic events in the prior 12 months or thromboembolic event of any grade with ongoing symptoms
6. Subjects with prior history of myocardial infarction, transient ischemic attack, congestive heart failure ≥ Class 3 based on New York Heart Association Functional Classification or stroke within the past 3 months prior to the scheduled first dose of study treatment
7. Active or prior documented autoimmune disorders within the past 3 years prior to the scheduled first dose of study treatment
8. HIV, Hep A, B, or C
9. History of primary immunodeficiency, solid organ transplantation, or active tuberculosis
10. Other invasive malignancy within 2 years
11. Known allergy or hypersensitivity to investigational product formulations
12. History of more than one event of infusion related reactions (IRR) requiring permanent discontinuation of IV drug treatment
13. Active grade 3 or greater edema
14. Uncontrolled intercurrent illness
15. Any history of leptomeningeal disease or cord compression
16. Untreated CNS metastatic disease.
17. Current or prior use of immunosuppressive medication within 14 days prior to the scheduled first dose of study treatment.
18. Receipt of live, attenuated vaccine within 30 days prior to the scheduled first dose of study treatment
19. Major surgery within 28 days prior to scheduled first dose of study treatment or still recovering from prior surgery
20. Females who are pregnant, lactating, or intend to become pregnant during their participation in the study
21. Subjects who are involuntarily incarcerated or are unable to willingly provide consent or are unable to comply with the protocol procedures
22. Any condition that, in the opinion of the investigator, would interfere with safe administration or evaluation of the investigational products or interpretation of subject safety or study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
cfMeDIP-seq-based assays of blood samples collected serially on study. Association between cfMeDIP and Toxicity (defined as ≥ Grade 2 immune- adverse event (AE) as per CTCAE 5.0) | 2 years
  Identify cfMeDIP-seq-based predictive signature(s) that are correlated with specific outcome to durvalumab and oleclumab such as response/resistance or occurrence of toxicity in pancreatic ductal adenocarcinoma (PDAC), non-small-cell carcinoma (NSCLC) and squamous cell carcinoma of head and neck (SCCHN).
Objective response rate (ORR) according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 | 2 years
Disease control rate (DCR) according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 | 2 years
Duration of response (DoR) | 2 years

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events (AEs) | 2 years
  To assess the safety and tolerability of durvalumab and oleclumab in specific disease states in PDAC, NSCLC and SCCHN
Overall survival (OS) | 2 years
Relapse-free survival (RFS) | 2 years
Progression-free survival (PFS) | 2 years
Pathological response rate in "Window" cohorts | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Lillian Siu, MD, Principal Investigator — Princess Margaret Cancer Centre
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No